CLINICAL TRIAL: NCT04602585
Title: The Effect of Psycho-education on Clinical Outcomes Among Patients With a First Episode Psychosis in Central Uganda - A Pilot Randomized Control Trial
Brief Title: The Effect of Psycho-education on Clinical Outcomes Among Patients With a First Episode Psychosis in Central Uganda
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Makerere University (Other)
Responsible Party: Principal Investigator, College of Health Sciences, Dr Dickens Akena, Makerere University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Psycho-education and Psychosis
Record Dates: First submitted 2020-10-20; First posted 2020-10-26 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Psychosis
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of 2 arms. There will be no cross over
Masking Description: We will mask participants at the point of randomization. They will pick a piece of paper that dictates which arm they will belong
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): After discharge, the program manager will link the participants with a VHT nearest to them. The participants (randomized to the intervention arm) will be informed during the consent procedure that they will undergo 6 psycho-education sessions (1 per month) together with a family member at the participant's residence. The VHTs and participants will meet and schedule appointments for the next engagements. This shall be done on a case by case basis. Some psycho-education sessions could take place in the patient's residence, others in the nearest public space (school or church or mosque compounds). The investigators will document where the majority of these sessions happen. This will help the investigators document feasibility. The PI and RAs will sit in some of the sessions during the pilot phase of data collection to ensure fidelity to the manual.
  Interventions: Behavioral: Psycho-education
- Usual care arm (Placebo Comparator): Participants will receive usual care
  Interventions: Behavioral: Psycho-education

INTERVENTIONS:
Behavioral: Psycho-education — Participants will receive 6 psycho-education sessions as adjunct therapy to the use of antipsychotics

SUMMARY:
Background: Psychotic disorders which the investigators have operationally defined as any of schizophrenia or schizophrenia spectrum disorder, brief psychotic episode, or bipolar affective disorders are severe forms of mental illness that contribute to significant morbidity and mortality primarily due to high rates of relapse. Delivering psycho-education messages about disease etiology, their signs and symptoms, as well as the benefits of adhering to treatment have been shown to reduce relapse among individuals with psychoses in high income countries. However, little has been done to examine the efficacy of this intervention in low resourced settings like Uganda.

Objective: The study objective is to examine the efficacy of psycho-education on symptom severity, stigma and retention in care.

Methods: The Investigators will recruit 80 adult patients (aged ≥18 years) who have been diagnosed with a First Episode Psychosis (FEP) and received antipsychotic medication at Butabika Hospital. Participants should be ready for discharge and reside within a 21km radius from Kampala city. The investigators will use a simple random technique to randomize the 80 participants to either receive 6 sessions of psycho-education from village health team members (VHTs) with a family member (n=40) or routine care (n=40). The investigators will collect symptom severity, stigma and retention in care data over 24 weeks.

Data analysis plans: The investigators will conduct an intention to treat analysis and compare the groups at baseline, weeks 4, 12 and 24. We will assess the effects of the intervention on symptom severity. The investigators will assess for potential confounders, mediators and effect modifiers using generalized linear estimates. Between-subject analysis at week 24 will be used to assess if there is a significant difference in the mean severity scores between the 2 arms.

Conclusion: Findings from this research will throw more light with regards to the preliminary efficacy of the use of psycho-education for individuals with psychosis.

DETAILED DESCRIPTION:
Methods

1. Study setting: The study will be conducted at the Butabika National Mental Referral Hospital in Kampala, a 600 bed hospital located 13km east of Kampala city
2. Eligibility criteria: Individuals will be eligible if they have been diagnosed with a First Episode Psychosis ( FEP) and considered (by the attending health care practitioner) to have demonstrable resolution of active symptoms following the use of antipsychotic medications, and deemed clinically stable for a discharge. The diagnosis of FEP will be confirmed through an interview conducted a by a research assistant (RA) using the Mini International Neuropsychiatric Instrument (MINI). Participants (adults ≥18 years) will be required to provide written informed consent and should reside within a 21 km radius from Kampala.

   Exclusion criteria: Individuals will be excluded if they present with a psychosis secondary to a medical or substance use disorder.
3. Sample size and power calculation: The investigators calculated the size of effects that our sample will be able to detect a clinically significant difference in symptom severity (primary outcome) between the two arms. A sample size of 80 (n=40 per arm) will provide sufficient power to detect a 50% difference in mean symptom severity levels between the two arms using a two-tailed z-test of proportions with 80% power and 95% confidence interval. Whereas this study is not adequately powered to detect statistical significance, our findings will provide the investigators with an effect size that can be used in sample size calculation of a powered randomized control trial (RCT).
4. Data collection methods

i) Training: RAs and VHTs will each undergo 4-day's training in the study procedures.

ii) Random sequence allocation: The investigators will use a simple random technique to randomize participants. Our biostatistician will write the words intervention, insert them in 40 opaque envelops and seal them, then do the same for controls

iii) Data collection: RAs shall identify potential participants, provide them with information about the study, obtain written informed consent, then administer the University of California, San Diego Brief Assessment of Capacity to Consent (UBACC) [40] to assess participant comprehension of the consent process.

RA's will administer a) standardized questionnaire to collect demographic and clinical variables (age, gender, address, education, date of symptom onset) b) MINI to confirm a diagnosis, c) Young Mania Rating Scale (YMRS) [41] for individuals with bipolar illness or Positive and Negative Symptoms of Schizophrenia Scale (PANSS) [42] for individuals with schizophrenia spectrum disorders to assess symptom severity d) World Health Organization Disability Assessment Schedule, e) Internalized Stigma of Mental Illness scale and f) a medication adherence measure

iv) Blinding participants and RA to the study arm: Participants will then pick an envelope and open it to see which study arm they belong. VHTs will deliver 6 psycho-education sessions (1 per month) to participants in intervention arm and their family members at the participant's residence. The PI and RAs will sit in some of the sessions during the pilot phase of data collection to ensure fidelity to the manual. RA's will schedule participants from both arms for an assessment using the same instruments at weeks 4, 12 and 24 at the clinic

v) Data analysis plans: The investigators will conduct an intention to treat analysis and compare the groups at baseline, weeks 4, 12 and 24. The investigators will assess the effects of the intervention on symptom severity (PANSS or YMRS). The investigators will assess for potential confounders, mediators and effect modifiers using generalized linear estimates.

Participant identification and recruitment:

i) Identification: Health care workers in the different wards and out-patient departments of Butabika Hospital will be informed about the study. Trained RA shall liaise with the clinicians to identify potential participants for recruitment at the time of admission to the wards. RA's will then assess participants who are due for discharge (patients with a clinical response to medications) for possible enrollment, and provide them with information about the study. Patients who access care at the out-patient clinic (who may not be admitted) but are eligible will also be approached by the RA for enrollment.

ii) The informed consent procedure: The RA's will invite potential participants to take part in the study, and obtain written informed consent. During the consenting process, the purpose of the study will be described further, the procedures will be explained, and the benefits of taking part in the study will be outlined. Upon demonstrating understanding and being given a chance to ask questions, the potential participant will then provide a witnessed, signed or thumb print consent.

iii) Assessing the capacity to consent: The investigators will administer the University of California, San Diego Brief Assessment of Capacity to Consent (UBACC) [40] instrument to assess whether the participants have understood the consent process. The UBACC will be translated into Luganda, the commonly spoken local language at the study site. The UBACC is a 10-item scale comprised of 3 factors that evaluate understanding, appreciation and reasoning. It has been used in the Ugandan setting for the Neuro-Genetics of Psychosis in African Populations (Neuro-GAP) project, although it is yet to be culturally adapted for use in these settings. A score of less than 14.5 on three separate occasions indicates that the participant has not understood what the study is all about. Such participants will not be recruited, but will be given a chance to return at a later date for recruitment (within a week). The investigators will record the number of participants who fail the UBACC at baseline and can't be recruited and those who do so after being invited a week later.

The investigators will ask participants to provide the investigators with their demographic information (age, gender and education level) and examine whether there are significant differences between participants who are able to consent and those who are not. Participation in this study is completely voluntary. The patient has the right to withdraw at any time during the study, including at follow-up. The investigators will document the reasons for withdrawal. Each interview is anticipated to last a minimum of 120 minutes -there will be 2-3 breaks at 40 minute intervals in between the interviews.

Feasibility of recruitment and delivery of care: The investigators anticipate recruiting the participants within 6 months. Since The investigators will recruit participants from the convalescent wards, they will administer the instruments over a 2 day period by conducting the consenting process a day earlier (takes approximately 30-45min). The rest of the interview will take approximately an hour and 15min. This is meant to reduce the time taken during the interviews. Furthermore, not all instruments will be administered in the same setting

1. The UBACC, Consent MINI, rating scales will be administered at baseline
2. At follow-up, The investigators will administer the MINI, rating scale, Medication adherence side rating scale (MARS) and WHO-disability adjusted life year scale (WHODAS). If the patient has Schizophrenia, they only get the PANSS and not the YMRS administered to them while if they have bipolar, they get the YMRS and not PNASS).

With each village having at least 5 VHTs, The investigators are confident that the participants will have access to at least one VHT within a 5km radius. The VHTs already play an integral part of ministry of health efforts including delivery of information during health campaigns as well as distribution of mosquito nets among many tasks initiated by the ministry. However, not all of them have received training in delivering mental health care. The investigators will identify them and train them.

ELIGIBILITY:
Inclusion Criteria:

* individuals will be eligible if they have been diagnosed with a FEP and considered (by the attending health care practitioner) to have demonstrable resolution of active symptoms following the use of antipsychotic medications, and deemed clinically stable for a discharge. The diagnosis of FEP will be confirmed through an interview conducted a by a research assistant (RA) using the Mini International Neuropsychiatric Instrument (M.I.N.I). Participants (adults ≥18 years) will be required to provide written informed consent and should reside within a 21 km radius from Kampala.

Exclusion Criteria:

* individuals will be excluded if they present with a psychosis secondary to a medical or substance use disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Reduction in symptom severity | 6 Months
  The investigators will measure a reduction in symptom severity as measured by the PANSS or YMRS

REFERENCES:
- [Derived] Akena D, Semeere A, Kadama P, Mwesiga EK, Nakku J, Nakasujja N. Feasibility of conducting a pilot randomized control trial of a psycho-education intervention in patients with a first episode psychosis in Uganda-A study protocol. PLoS One. 2022 Jul 29;17(7):e0268493. doi: 10.1371/journal.pone.0268493. eCollection 2022. PMID 35905117